CLINICAL TRIAL: NCT00063635
Title: Clinical Research Network in Nonalcoholic Steatohepatitis: Treatment of Nonalcoholic Fatty Liver Disease in Children (TONIC)
Brief Title: Treatment of Nonalcoholic Fatty Liver Disease in Children (TONIC)
Acronym: TONIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NASH - PEDIATRICS (IND)
Record Dates: First submitted 2003-07-01; First posted 2003-07-03 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-08

CONDITIONS: Fatty Liver
Keywords: Non alcoholic fatty liver disease
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Metformin; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Metformin, 500 mg, twice daily
  Interventions: Drug: Metformin
- 2 (Active Comparator): Vitamin E, 400 IU, twice daily
  Interventions: Dietary Supplement: Vitamin E
- 3 (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Metformin — 500 mg, twice daily
  Arms: 1
Dietary Supplement: Vitamin E — 400 IU, twice daily
  Other Names: Nature Made
  Arms: 2
Drug: Matching placebo — Twice daily
  Arms: 3

SUMMARY:
The purpose of this study is to determine if therapeutic modification of insulin resistance or oxidative stress leads to improvement in serum or histologic indicators of liver injury or quality of life.

ELIGIBILITY:
* Age 8-17 years at first screening visit
* Histologic evidence of Nonalcoholic Fatty Liver Disease (NAFLD) - biopsy cannot be older than 6 months as of randomization
* ALT level >60 U/L at time of screening and on one previous occasion determined at least one month but no greater than 6 months prior to screening ALT
* Consent

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - St. Louis University, St Louis, Missouri
  - Case Western Reserve University, Cleveland, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Corey KE, Vuppalanchi R, Vos M, Kohli R, Molleston JP, Wilson L, Unalp-Arida A, Cummings OW, Lavine JE, Chalasani N; Nonalcoholic Steatohepatitis Clinical Research Network. Improvement in liver histology is associated with reduction in dyslipidemia in children with nonalcoholic fatty liver disease. J Pediatr Gastroenterol Nutr. 2015 Mar;60(3):360-7. doi: 10.1097/MPG.0000000000000584. PMID 25714579
- [Derived] Guerrerio AL, Colvin RM, Schwartz AK, Molleston JP, Murray KF, Diehl A, Mohan P, Schwimmer JB, Lavine JE, Torbenson MS, Scheimann AO. Choline intake in a large cohort of patients with nonalcoholic fatty liver disease. Am J Clin Nutr. 2012 Apr;95(4):892-900. doi: 10.3945/ajcn.111.020156. Epub 2012 Feb 15. PMID 22338037
- [Derived] Lavine JE, Schwimmer JB, Van Natta ML, Molleston JP, Murray KF, Rosenthal P, Abrams SH, Scheimann AO, Sanyal AJ, Chalasani N, Tonascia J, Unalp A, Clark JM, Brunt EM, Kleiner DE, Hoofnagle JH, Robuck PR; Nonalcoholic Steatohepatitis Clinical Research Network. Effect of vitamin E or metformin for treatment of nonalcoholic fatty liver disease in children and adolescents: the TONIC randomized controlled trial. JAMA. 2011 Apr 27;305(16):1659-68. doi: 10.1001/jama.2011.520. PMID 21521847
- [Derived] Lavine JE, Schwimmer JB, Molleston JP, Scheimann AO, Murray KF, Abrams SH, Rosenthal P, Sanyal AJ, Robuck PR, Brunt EM, Unalp A, Tonascia J; Nonalcoholic Steatohepatitis Clinical Research Network Research Group. Treatment of nonalcoholic fatty liver disease in children: TONIC trial design. Contemp Clin Trials. 2010 Jan;31(1):62-70. doi: 10.1016/j.cct.2009.09.001. Epub 2009 Sep 15. PMID 19761871
- See also: National Institute of Diabetes and Digestive and Kidney Diseases — http://www.niddk.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2005 and September 2007, 173 children were enrolled into TONIC at 10 clinical centers in the United States.
Groups:
- Metformin: Metformin, 500 mg, twice daily
- Vitamin E: Vitamin E, 400 IU, twice daily
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | Metformin | Vitamin E | Placebo
Started | 57 | 58 | 58
Completed | 51 | 50 | 49
Not Completed | 6 | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Vitamin E | Placebo | Total
Number analyzed (Participants) | 57 | 58 | 58 | 173
Age Continuous [Mean (Standard Deviation); unit: years] | 13.1 (2.4) | 13.4 (2.3) | 12.9 (2.6) | 13.1 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 12 | 33
  Male | 47 | 47 | 46 | 140
Region of Enrollment [Number; unit: participants]
  United States | 57 | 58 | 58 | 173
NAFLD activity score [Mean (Standard Deviation); unit: scores on a scale] — Total nonalcoholic fatty liver disease (NAFLD) activity was assessed on a scale of 0 to 8, with higher scores indicating more severe disease; the components of this measure include steatosis (assessed on a scale of 0 to 3), lobular inflammation (assessed on a scale of 0 to 3), and hepatocellular ballooning (assessed on a scale of 0 to 2).
  scores on a scale | 4.5 (1.2) | 4.8 (1.6) | 4.6 (1.3) | 4.6 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Reduction in Alanine Aminotransferase (ALT) to Either 50% of Baseline Value or < 40 IU/L
Description: The primary outcome was sustained reduction in ALT level, defined as 50% or less of the baseline level or 40 IU/L or less at each visit from 48 to 96 weeks of treatment.
Time Frame: baseline and 96 weeks
Population: All enrolled patients were included in analysis of the primary outcome, sustained reduction in ALT level. Patients missing a 96-week ALT measurement were imputed as not achieving a sustained reduction.
Measure: Number; unit: participants
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 57 | 58 | 58
participants | 9 [7 to 28] | 15 [15 to 39] | 10 [9 to 29]
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.26, Mantel Haenszel — Since two primary comparisons are planned, a P-value of 0.025 will be considered significant, applying a Bonferroni correction for multiple comparisons
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.83, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Serum Aspartate Aminotransferase (AST)
Time Frame: baseline and 96 weeks
Measure: Mean (95% Confidence Interval); unit: IU/L
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 51 | 50 | 49
IU/L | -21.5 [-34.6 to -8.4] | -22.8 [-33.3 to -12.3] | -20.4 [-32.7 to -8.0]
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.32, ANCOVA
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.29, ANCOVA

3. Secondary Outcome: Change in Nonalcoholic Fatty Liver Disease (NAFLD) Score (Histologic Feature Scores Determined by Standardized Scoring of Liver Biopsies) From Baseline at 96 Weeks of Treatment
Description: Histological activity was assessed using the NAFLD activity score on a scale of 0 to 8, with higher scores indicating more severe disease; the components of this measure include steatosis (0-3), lobular inflammation (0-3), and hepatocellular ballooning (0-2).
Time Frame: baseline and 96 weeks
Population: Number of participants analyzed reflects the number of participants with baseline and 96 week liver biopsies.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 50 | 50 | 47
units on a scale | -1.1 [-1.7 to -0.5] | -1.8 [-2.4 to -1.2] | -0.7 [-1.3 to -0.2]
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.02, ANCOVA
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.25, ANCOVA

4. Secondary Outcome: Number of Participants With Improvement in Liver Fibrosis Score
Description: Fibrosis is assessed on a scale of 0 to 4 with higher scores indicating more severe fibrosis. This secondary outcome measure is the number of participants that experienced a decrease in fibrosis score at 96 weeks compared to baseline, which indicates improvement in fibrosis.
Time Frame: baseline and 96 weeks
Population: Number of participants analyzed reflects the number of participants with baseline and 96 week liver biopsies.
Measure: Number; unit: participants
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 50 | 50 | 47
participants | 22 | 18 | 19
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.71, Chi-squared
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.72, Chi-squared

5. Secondary Outcome: Number of Participants With Improvement in Steatosis Score
Description: Steatosis is assessed on a scale of 0 to 3 with higher scores indicating more severe steatosis. This secondary outcome measure is the number of participants that experienced a decrease in steatosis score at 96 weeks compared to baseline, which indicates improvement in steatosis.
Time Frame: baseline and 96 weeks
Population: Number of participants analyzed reflects the number of participants with baseline and 96 week liver biopsies.
Measure: Number; unit: participants
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 50 | 50 | 47
participants | 26 | 27 | 19
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.18, Chi-squared
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.25, Chi-squared

6. Secondary Outcome: Number of Participants With Improvement in Lobular Inflammation Score
Description: Lobular inflammation is assessed on a scale of 0 to 3 with higher scores indicating more severe lobular inflammation. This secondary outcome measure is the number of participants that experienced a decrease in lobular inflammation score at 96 weeks compared to baseline, which indicates improvement in lobular inflammation.
Time Frame: baseline and 96 weeks
Population: Number of participants analyzed reflects the number of participants with baseline and 96 week liver biopsies.
Measure: Number; unit: participants
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 50 | 50 | 47
participants | 23 | 22 | 20
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.89, Chi-squared
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.73, Chi-squared

7. Secondary Outcome: Number of Participants With Improvement in Ballooning Degradation Score
Description: Ballooning is assessed on a scale of 0 to 2 with higher scores indicating more severe ballooning. This secondary outcome measure is the number of participants that experienced a decrease in ballooning score at 96 weeks compared to baseline, which indicates improvement in ballooning.
Time Frame: baseline and 96 weeks
Population: Number of participants analyzed reflects the number of participants with baseline and 96 week liver biopsies.
Measure: Number; unit: participants
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 50 | 50 | 47
participants | 22 | 22 | 10
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.02, Chi-squared
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.02, Chi-squared

8. Secondary Outcome: Change in Body Mass Index
Time Frame: baseline and 96 weeks
Measure: Mean (95% Confidence Interval); unit: kg/m-squared
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 51 | 50 | 49
kg/m-squared | 1.3 [0.6 to 2.0] | 2.1 [1.2 to 3.0] | 1.9 [1.1 to 2.7]
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.77, ANCOVA
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.25, ANCOVA

9. Secondary Outcome: Change in Serum Vitamin E Levels
Description: Change in alpha-Tocopherol
Time Frame: baseline and 96 weeks
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 51 | 50 | 49
mg/L | -0.5 [-1.1 to 0.2] | 9.4 [6.2 to 12.6] | -0.9 [-2.1 to 0.4]
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.44, ANCOVA

10. Secondary Outcome: Change in Quality of Life (QOL) Scores- Physical Health
Description: Change in self-reported QOL physical health Pediatric Quality of Life Inventory (version 4.0) scores were recorded to range from 0 to 100 with increasing scores indicating better quality of life.
Time Frame: baseline and 96 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 51 | 50 | 49
units on a scale | 5.4 [0.8 to 10.0] | 7.6 [2.7 to 12.5] | 5.4 [-0.7 to 11.5]
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.08, ANCOVA
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.63, ANCOVA

11. Secondary Outcome: Change in QOL- Psychosocial Health
Description: as for outcome 10
Time Frame: baseline and 96 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Metformin | Vitamin E | Placebo
Number analyzed (Participants) | 51 | 50 | 47
units on a scale | 4.0 [-0.4 to 8.4] | 6.0 [1.4 to 10.6] | 5.6 [0.0 to 11.2]
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.15, ANCOVA
Statistical Analysis 2: Comparison: Metformin vs Placebo; Test type: Superiority or Other; p = 0.96, ANCOVA

ADVERSE EVENTS:
Arm/Group | Metformin | Vitamin E | Placebo
Serious Adverse Events (participants affected / at risk) | 7/57 | 6/58 | 14/58
Other Adverse Events (participants affected / at risk) | 17/57 | 17/58 | 18/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=57) | Vitamin E (N=58) | Placebo (N=58)
Airway constriction/bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Appendicitis (Gastrointestinal disorders) | 1 | 0 | 1
Cholecystitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (General disorders) | 1 | 0 | 0
Diabetes (Endocrine disorders) | 0 | 0 | 1
Elevated serum glucose (Endocrine disorders) | 1 | 1 | 0
Hepatobiliary/pancreas (Hepatobiliary disorders) | 0 | 0 | 5
Hepatotoxicity (Hepatobiliary disorders) | 2 | 1 | 0
Pain (General disorders) | 1 | 0 | 1
Syncope (Cardiac disorders) | 0 | 1 | 1
(General disorders) | 0 | 0 | 1
Depression (General disorders) | 1 | 1 | 2
Suicide (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=57) | Vitamin E (N=58) | Placebo (N=58)
Unspecified- Mild (General disorders) | 10 | 10 | 6
Unspecified- Moderate (General disorders) | 7 | 7 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No